CLINICAL TRIAL: NCT01318187
Title: Intravenous Paracetamol or Morphine for the Treatment of Acute Flank Pain : a Randomized, Double Blind, Controlled Clinical Trial
Brief Title: Intravenous Paracetamol or Morphine for the Treatment of Acute Flank Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: serinken 001
Record Dates: First submitted 2011-03-17; First posted 2011-03-18 (Estimated); Last update posted 2011-04-01 (Estimated); Status verified 2011-01

CONDITIONS: Urolithiasis
Keywords: renal colic; paracetamol; morphine; emergency department
MeSH Terms: conditions — Urolithiasis; Renal Colic; Emergencies | interventions — Acetaminophen; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paracetamol (Experimental)
  Interventions: Drug: paracetamol; Drug: morphine
- Morphine (Active Comparator)
  Interventions: Drug: paracetamol; Drug: morphine

INTERVENTIONS:
Drug: paracetamol — 1 gr
  Other Names: Perfalgan
Drug: morphine — 0.1mg/kg intravenous in 100 ml serum physiologic
  Other Names: Morphine CHL 0.01 gr
Drug: Paracetamol — 1 gr intravenous
  Other Names: Perfalgan
  Arms: Paracetamol
Drug: Paracetamol — intravenous 1 gr
  Other Names: Perfalgan
  Arms: Paracetamol
Drug: Morphine — 0.1 mg/kg intravenous
  Arms: Morphine

SUMMARY:
STUDY OBJECTIVE: This randomized, controlled trial evaluates the analgesic efficacy and safety of intravenous single-dose paracetamol and morphine for the treatment of acute flank pain.

METHODS: The investigators conducted a randomized, double-blind, controlled clinical trial comparing single intravenous doses of paracetamol (1 g) and morphine (0.1 mg/kg) for patients presenting to the emergency department (ED) with acute flank pain. Subjects with inadequate pain relief at 30 minutes received rescue fentanyl (0.75 microg/kg).

DETAILED DESCRIPTION:
Study Design and Setting:

This is a single-center, prospective, randomized, double-blind, clinical trial performed in an ED of a tertiary care hospital with annual census of approximately 37.000 visits. The local ethics committee approved the study.

Two treatment options, intravenous paracetamol and morphine, were compared for ceasing pain in patients presented with renal colic.

Selection of Participants:

Patients, aged 18 to 55 years, with flank pain were accepted as eligible for the study. Patients with clinical diagnosis of acute renal colic and declared to have moderate or serious pain according to the 4-point verbal scale were included into the study.

Exclusion criteria were as follows: patients denied to give inform consent, use of any analgesic within six hours of ED presentation, patients with fewer or hemodynamically unstable, peritoneal irritation signs, cardiac failure, history of renal and hepatic failure, prior known allergy to paracetamol or morphine, suspected or documented pregnancy and patients with viewing problems. Patients suspected to have renal colic but ultimately to have diagnosis such as renal abscess, renal infarction or renal venous thrombosis were also excluded from the study.

Consecutive patients were enrolled into the study 24 hours a day and seven days a week by the senior resident in the shift. The ultimate diagnosis of renal colic was performed by displaying the stone either by ultrasonograph (USG) or computerized tomography (CT). USG was the first choice for detecting the renal stone. CT was performed if a stone was not detected by USG. After CT, patients who were not shown a urolithiasis or pathologies other than renal colic were excluded from the study.

Interventions:

Study subjects were randomized in order to receive a single dose of either paracetamol (Perfalgan, Bristol Myers Squibb, Itxassou, France), 1 gr in 100 ml normal saline, or morphine (0.1 mg/kg in 100 ml normal saline) in a blinded fashion. The study drugs was written in a paper which is folded four times and covered with sealed bands for allocation concealment. The study nurse withdrew one of the drugs from a box. And they were prepared by the study nurse and administered by the second nurse blinded to the study. Study drugs were identical in color and appearance. Subjects with who needed rescue drug because of inadequate pain relief were received fentanyl 1 μg/kg intravenously.

Methods of Measurements:

Subjects reported pain intensity on both a 100-mm visual analogue scale (limited by 'no pain' and 'the worst pain') and a 4-point verbal rating scale (no pain, mild, moderate, or severe pain) just before the drug administration, 15th minutes and 30th minutes after the study drug administration. The demographic features of study patients and adverse effects, nausea, vomiting, dizziness, vertigo, headache, hypotension, altered mental status, allergic reaction, itching, urinary retention, thoracic rigidity, respiratory depression and dry mouth, were recorded to the study form.

Outcome Measures The primary outcome measure was the pain reduction in VAS and VRS at 15th and 30th minutes. Secondary outcome measures were the need for rescue drug and the presence of any adverse event.

Primary Data Analysis:

The present study was planned as a superiority trial. When the 20 mm difference in VAS is accepted as clinically significant and the standard deviation is accepted as 25 mm, 35 patients are needed with each group with 95% power. All the analysis were implemented according to the intention to treat analysis. The precise of differences between time intervals within groups and between groups and statistical significance were expressed by 95% confidence intervals (95% CI). All tests of significance were two sided.

ELIGIBILITY:
Inclusion Criteria:

Adults (aged 16 to 55 years old) with acute low back pain were eligible for inclusion in the study

Exclusion Criteria:

* known allergy or contraindication to morphine, paracetamol, or any opioid analgesic
* hemodynamic instability; fever (temperature > 38°C [100.4°F])
* evidence of peritoneal inflammation
* documented or suspected pregnancy
* known or suspected aortic dissection or aneurysm
* use of any analgesic within 6 hours of ED presentation
* previous study enrollment Patients with known renal, pulmonary, cardiac, or hepatic failure, as well as those with renal transplantation, were also excluded.

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 73 (Actual)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Reduction in visual analogue scale | 15 minutes interval
  The pain of the study subjects was measured after 15th and 30th minutes later after the study drug administered.

SECONDARY OUTCOMES:
Adverse events. | 30th minutes after
  30th minutes after the study drug administered

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Serinken, Proffesor, Study Director — Pamukkale University
Locations (2):
- Turkey (Türkiye) (2):
  - Pamukkale University Hospital Emergency Department, Denizli
  - Pamukkale University, Denizli

REFERENCES:
- [Result] Bektas F, Eken C, Karadeniz O, Goksu E, Cubuk M, Cete Y. Intravenous paracetamol or morphine for the treatment of renal colic: a randomized, placebo-controlled trial. Ann Emerg Med. 2009 Oct;54(4):568-74. doi: 10.1016/j.annemergmed.2009.06.501. Epub 2009 Jul 31. PMID 19647342
- [Derived] Serinken M, Eken C, Turkcuer I, Elicabuk H, Uyanik E, Schultz CH. Intravenous paracetamol versus morphine for renal colic in the emergency department: a randomised double-blind controlled trial. Emerg Med J. 2012 Nov;29(11):902-5. doi: 10.1136/emermed-2011-200165. Epub 2011 Dec 20. PMID 22186009